CLINICAL TRIAL: NCT05426811
Title: Regorafenib Plus Raltitrexed as Third-line Treatment in Advanced Colorectal Cancer Patients：An Open-label, Single-arm, Multicenter Phase I/II Study
Brief Title: Regorafenib Plus Raltitrexed as Third-line Treatment in Advanced Colorectal Cancer Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University, China (Other)
Collaborators: The People's Hospital of Liaoning Province (Other); Anshan Tumor Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Benxi Cental Hospital (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, Director of Department of Medical Oncology, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REGORAL
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Regorafenib; Raltitrexed; Colorectal Neoplasms; Third-line Treatment
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib; raltitrexed

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regorafenib combined with Raltitrexed (Experimental): Regorafenib:
  120mg/d，Po，qd,d1-d21，Every 4 weeks
  Raltitrexed:
  3mg/㎡，ivgtt，d1，Every 3 weeks
  Interventions: Drug: Regorafenib; Drug: Raltitrexed

INTERVENTIONS:
Drug: Regorafenib — Regorafenib:120mg/d，Po，qd,d1-d21，Every 4 weeks
  Other Names: Stivarga
Drug: Raltitrexed — Raltitrexed:3mg/㎡，ivgtt，d1，Every 3 weeks
  Other Names: Sai wei jian

SUMMARY:
This is a multicenter, open, single-arm, phase I/II study to evaluate the efficacy and safety of regorafenib plus raltitrexed as third-line treatment in patients with advanced colorectal cancer.

DETAILED DESCRIPTION:
This is a multicenter, open, single-arm, phase I/II study to evaluate the efficacy and safety of regorafenib plus raltitrexed as third-line treatment in patients with advanced colorectal cancer.This Phase Ib/II study consists of two parts, Phase Ib, an open-ended, single-arm, multi-centre, dose-escalation study evaluating regorafenib, and Phase II, an open-label, multi-centre study evaluating the efficacy and safety of regorafenib in combination with raltitrexed.The primary study endpoint: progression-free survival (PFS).The secondary end endpoints include ORR (overall effectiveness of tumour treatment)，DCR (disease control rate)，3 month/6 month/9 month/12 month survival OS%，OS (overall survival)，incidence and severity of adverse events (AEs), serious adverse events (SAEs).

ELIGIBILITY:
Inclusion Criteria

1. Sign a consent form
2. Age> 18 years
3. Pathological diagnosis as metastatic colorectal adenocarcinoma
4. Metastatic colorectal cancer with disease progression after 1st and 2nd line treatment；Received standard chemotherapy based on fluorouracil, oxaliplatin, irinotecan, patients are allowed to receive EGFR and/or VEGF inhibitors, patients are allowed to receive immunotherapy.
5. Measurable disease according to RECIST
6. ECOG score 0-1 points
7. Life expectancy ≥3 months
8. ALT and AST< 2.5 times the upper limit of normal (ULN), patients with liver metastases < 5 times ULN
9. Serum albumin ≥ 3.0g/ dL
10. Serum ALP <2.5 times ULN
11. Total bilirubin <l.5mg / dL
12. Estimated creatinine clearance (CLcr) ≥30mL/min as calculated using the Cockcroft-Gault equation
13. Lipase≤1.5x the ULN
14. Neutrophil absolute count (ANC) ≥1500/mm³, hemoglobin (Hb)>9g/dl, platelets> 10000/mm³
15. Pregnant or breastfeeding patients. (1) Women and men of childbearing potential must agree to use appropriate contraception prior to entering the program until at least 8 weeks after the last dose of study drug. The investigator or designee is required to advise the subject on how to achieve appropriate contraception. Adequate contraception is defined in the study as any medically recommended method (or combination of methods) according to standard treatment 2) Women of childbearing age must confirm a negative serum or urine pregnancy test within 7 days prior to initiating treatment and must agree to record a negative result prior to entering the study

Exclusion criteria.

1. Prior exposure to any VEGFR tyrosine kinase inhibitor (e.g., regorafenib, apatinib, anlotinib, furoquinitinib, etc.) therapy
2. Received raltitrexed in the previous treatment
3. Patients with abnormal coagulation function or those treated with thrombolytic or anticoagulant drugs with a tendency to bleed from the gastrointestinal tract, including active peptic ulcer with fecal occult blood ++, vomiting blood or black stool within 3 months
4. Prior or concurrent cancers with a different primary site or histology than CRC within the enrollment year, except cured in situ cervical cancer, non-melanoma skin cancer, and superficial bladder tumors: staged Ta, Tis, and T1
5. Arterial or venous thrombotic or embolic events such ascerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 month before the start of study medication (except for adequately treated catheter-related venous thrombos is occurring more than one month before the start of study medication)
6. Major surgery, biopsy or significant traumatic damage within 28 days prior to the start of investigational treatment
7. Non-healing wound, non-healing ulcer, or non-healing bone fracture.
8. Patients with brain metastases and/or cancerous meningitis
9. Congestive heart failure > New York Heart Association (NYHA) class 2.
10. Unstable angina (angina symptoms at rest), new onset angina (occurred within the last 3 months). Myocardial infarction within 6 months prior to the start of treatment.
11. Arrhythmias requiring antiarrhythmic therapy (beta-blockers or digoxin allowed)
12. Uncontrolled hypertension. (Systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg despite optimal medical treatment)
13. Patients with pheochromocytoma
14. Pleural effusion or ascites causing restricted breathing (≥ CTCAE grade 2 dyspnea)
15. Known to have dihydropyrimidine dehydrogenase deficiency
16. Ongoing infection > Grade 2 NCI CTCAE
17. Interstitial lung disease with ongoing signs and symptoms at the time of informed consent
18. Known hypersensitivity to any of the stidy drugs, study drug classes,or excipients in the formulation
19. The use of CYP3A4 inhibitors or inducers
20. Participation in another clinical trial within 4 weeks prior to enrollment and receipt of the investigational drug and any concomitant therapy containing the investigational drug
21. Received radiotherapy within 4 weeks prior to enrollment and the lesions observed in this study were in the target area of radiotherapy
22. Subjects with active tuberculosis (TB) who are on anti-tuberculosis treatment, or who have received anti-tuberculosis treatment within one year prior to screening
23. Comorbidities requiring long-term treatment with immunosuppressive drugs or systemic or topical corticosteroids at immunosuppressive doses (doses >10 mg/day of prednisone or other isotonic hormones)
24. Received any anti-infective vaccine (e.g., influenza vaccine, varicella vaccine, Neocon vaccine, etc.) within 4 weeks prior to enrollment
25. Pregnancy or breastfeeding
26. Persistent proteinuria >3.5g/24 hours by measuring the urine protein-creatinine ratio in random urine samples (grade 3, NCI-CTCAE version 5.0)
27. Positive for Human Immunodeficiency Virus (HIV)
28. Positive hepatitis B virus surface antigen (HBsAg) with positive HBV DNA copy number (quantitative test ≥ 1000 cps/ml)
29. Positive blood screen for chronic hepatitis C (positive for HCV antibodies)
30. Renal failure requiring hemodialysis or peritoneal dialysis
31. The degree of dehydration ≥ CTCAE version 5.0 level 1
32. Persons without legal capacity
33. Any other clinically significant disease or condition that, in the opinion of the investigator, could affect compliance with the protocol, or affect the subject's ability to sign an informed consent form (ICF), or is inappropriate for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | one year
  PFS, defined as the time from randomization to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | one year
  ORR, determined using RECIST v1.1, defined as best overall response (CR or PR) across all assessment time points during the period from enrolment to termination of trial treatment.
Disease Control Rate (DCR) | one year
  Determined using RECIST v1.1 criteria.
Overall Survival (OS) | two years
  Duration from the date of initial treatment to the date of death due to any cause.
Incidence and severity of adverse events (AE) and serious adverse events (SAE) | two years
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Liu, PhD, Principal Investigator — First Hospital of China Medical University

IPD SHARING:
Plan to Share IPD: No